CLINICAL TRIAL: NCT06399770
Title: The Role of Muscle Ultrasound in Assessment of Sample of Patients With Limb-girdle Muscular Dystrophy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Bassem Fikry Ramzy, Abanoub bassem, Assiut University
Other Study IDs: Limb-girdle muscular dystrophy
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Limb-girdle Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Muscle ultrasound — Role of muscle ultrasound in LGMD

SUMMARY:
1. to detect the characteristic patterns of muscle involvement in suspected cases of LGMD using muscle ultrasound
2. to use the muscle ultrasound findings clinically categorized the different types of LGMD
3. to correlate the muscle ultrasound findings with the findings of the other assissed scales

DETAILED DESCRIPTION:
Limb-girdle muscular dystrophies (LGMD) are muscular dystrophies that affect skeletal muscles, mostly proximal (hips and shoulder muscles). They are caused by a mutation in a gene encoding a protein, which is specific to each subtype. LGMD inheritance is either autosomal dominant or recessive. Several types of LGMD were described depending on the causative mutations (1). LGMD is one of inherited myopathies that characterized by selective involvement of muscles. Selectivity is a sign of muscle diseases and helps direct the diagnosis; however, it cannot always be identified clinically; consequently, the importance of using muscle MRI and ultrasound are to detect this selectivity and aid in the diagnosis (2). Ultrasound with a high resolution enables viewing of the muscle, nerve, and nearby structures and can provide real-time information in neuromuscular illnesses (3). Muscle Ultrasound (MUS) can detect the same patterns of muscle affection as MRI (4). In addition, it is safe, accessible, low-cost, and free of ionizing radiation, with no known contraindications and no difficulties associated with MRI, such as claustrophobia, metallic implants, and the requirement for sedation in children; hence, it can be used as a supplemental technique to electro- diagnosis (5). Ultrasound can provide real-time information related to muscle activation and movement patterns; so, selective substitution of muscle ultrasound for MRI can result in significant cost-saving for the health care system (6). However, its primary drawback is that it is operator-dependent and has a limited ability to image deeper structures (7). According to studies, MUS can provide a key provisional probable diagnosis, especially when genetic diagnosis is not accessible or expensive, or to provide guide to the proper genetic testing when it is available (2, 8). In limb girdle pattern of weakness patients, MUS assisted diagnose quadriceps sparing myopathy, selective affection of one head of gastrocnemius as medial head and soleus more than lateral head in FKRP (LGMD2I) and calpain-3 deficiency (LGMD2A), and selective affection of lateral head as in LGMD2B.

(dysferlin) (9). MUS can also help diagnose the treatable types of limb girdle myopathies like POPME by recognizing specific muscle involvement patterns (2). Few research (10), utilized the MUS to detect suspected LGMD, and none compared the MUS findings with those of the different psychometric measures. The present study aims to we aimed to evaluate the role of MUS in the assessment of patients with suspected LGMD to identify characteristic patterns these of muscle involvement in suspected cases of LGMD and to correlate changes with findings of the different psychometric scales.

ELIGIBILITY:
Inclusion Criteria:

* gender : both sex are included Willingness to participate in the study and to be subjected to disease related examination and assessments Willing and able to provide informd consent

Exclusion Criteria:

* patients unable to give informed consent Patients with acute or subacute onset of symptoms of muscle involvement including inflammatory myopathies Patients with systemic diseases causing secondary myopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients presented with clinical manifestations suggestive of LGMD who presented with gradual progressive limb-girdle weakness ,myopathic changes on electromyography and elevated creatine phosphokinase serum level
  * age and sex matched healthy control group as a normal referencce
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The role of muscle ultrasound in assessment of a sample of patients with limb-girdle muscular dystrophy | Baseline
  The role of muscle ultrasound in assessment of sample of patients with LGMD